CLINICAL TRIAL: NCT01784380
Title: The Potential Biochemical Diagnosis Criteria and Therapeutic Effect Indexes: Sex Hormone Binding Globulin Levels and Free Androgen Index in Blood of Patients With Polycystic Ovary Syndrome
Status: Completed | Type: Observational
Sponsor: Zhongshan Bo Ai Hospital (Other)
Responsible Party: Principal Investigator, LIN Xiu-feng, physician, Zhongshan Bo Ai Hospital
Other Study IDs: 2006A165
Record Dates: First submitted 2013-01-30; First posted 2013-02-05 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-02

CONDITIONS: The Investigators Collected 534 PCOS Patients as the Case Group,and 580 Infertile Women With Normal Ovulatory Cycle of the Control Group;; At the Same Time, the Investigators Continuedly Collect Cases to October 2012, and Totally Collected 579 Patients With PCOS Altogether;; 534 Patients in the Cases Group and 580 Women in the Control Group Received no Measures, While 579 Patients Received Drugs;; The Investigators Monitored Basic Indexes in Blood of All the Subjects in This Suvey,and Also Monitored Indexes of 579 Patients After Treatment.
MeSH Terms: interventions — Menotropins

STUDY DESIGN:
Observational Model: Case-Control

GROUPS / COHORTS (3):
- the case group
- the control group
- the treatment group: Patients of the treatment group recieved drugs,then we observed drugs' treatment effect.
  Interventions: Drug: Diane-35;metformin;Clomiphene citrate; Human menopausal gonadotropin

INTERVENTIONS:
Drug: Diane-35;metformin;Clomiphene citrate; Human menopausal gonadotropin
  Groups: the treatment group

SUMMARY:
To explore whether Free androgen index（FAI）can be regarded as biochemically diagnostic indexes of high androgen hormone in blood of patients with Polycentric ovary syndrome（PCOS）. Also to explore whether Sex hormone-binding globulin（SHBG） and FAI can be seen as therapeutic effect indicatrixes of women with PCOS.

ELIGIBILITY:
Inclusion Criteria:

* The clinical diagnosis criteria for PCOS by European Society of Human Reproduction and Embryology, and Rotterdam working group of American Society for Reproductive Medicine (ESHRE /ASRM )

Exclusion Criteria:

* hyperprolactinemia and other endocrine diseases such as high androgen hormone in blood, namely Cushing's syndrome, congenital adrenal hyperplasia ( CAH ), ovarian or adrenal tumor and so on

Ages: 20 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The investigators collected 534 PCOS patients as the case group, 580 infertile women with normally ovulatory cycle as the control groupand.The patients of the case group aged from 20 to 42 years old, the average age was 27.87 years old, and the standard deviation of ages was 3.75 years old. And patients' ovulation in the case group was normal, as control group, aged from 20 to 43 years old, the average age was 28.18 years old; the standard deviation of ages was 3.99 years old.Also the investigators also collected 579 patients as the treatment group,who aged from 20 to 39 years, the average age was 27.93 years old, the standard deviation of ages was 3.70 years old.
Sampling Method: Probability Sample
Enrollment: 1159 (Actual)
Dates: Start 2006-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
The potentially biochemical diagnosis criteria and therapeutic effect evaluation indexes: Sex hormone binding globulin levels and free androgen index in blood of patients with polycystic ovary syndrome | after 5 weeks of ovulation treatment

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Elecsys2010,French KONTRON EUB-5500 color Doppler ultrasonic diagnostic apparatus, Zhongshan, Guangdong
  - Reproductive Center of Bo Ai Hospital, Zhongshan, Zhongshan, Guangdong

REFERENCES:
- [Result] Zolghadri J, Tavana Z, Kazerooni T, Soveid M, Taghieh M. Relationship between abnormal glucose tolerance test and history of previous recurrent miscarriages, and beneficial effect of metformin in these patients: a prospective clinical study. Fertil Steril. 2008 Sep;90(3):727-30. doi: 10.1016/j.fertnstert.2007.06.079. Epub 2007 Nov 14. PMID 18001723